CLINICAL TRIAL: NCT06581536
Title: Rigorous Evaluation of Yes and Know, a Fully Virtual Intervention Integrating Group-based Education With Digital Tools to Improve Youth Sexual Health and Well-Being
Brief Title: Rigorous Evaluation of Yes and Know, a Fully Virtual Sexual Health and Well-Being Intervention for Youth
Acronym: Yes and Know
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ETR Associates (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TP2AH000079
Record Dates: First submitted 2024-08-29; First posted 2024-09-03 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy Related; Sexually Transmitted Diseases; Adolescent Behavior
MeSH Terms: conditions — Sexually Transmitted Diseases; Adolescent Behavior | interventions — YES1 protein, human; Nutrition Assessment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yes and Know curriculum (Experimental): Youth will receive the Yes and Know curriculum.
  Interventions: Behavioral: Yes and Know curriculum
- Nutrition Education for Adolescents (Active Comparator): Youth will receive education about adolescent nutrition.
  Interventions: Behavioral: Nutrition Education for Adolescents

INTERVENTIONS:
Behavioral: Yes and Know curriculum — Yes and Know is fully virtual intervention that integrates group-based education with digital tools to support young people ages 14 to 19 by increasing their relationship and healthy life skills. The curriculum focuses on sexual and reproductive health; healthy relationships; life skills; and educational and career success. It is delivered over nine synchronous sessions of 60-minutes each for a duration of nine hours, plus asynchronous online resources and activities.
  Arms: Yes and Know curriculum
Behavioral: Nutrition Education for Adolescents — Youth will receive a fully virtual intervention that integrates group-based education with digital tools focused on adolescent nutrition and wellness. The curriculum is delivered over nine synchronous sessions of 60-minutes each for a duration of nine hours, plus asynchronous online resources and activities.
  Arms: Nutrition Education for Adolescents

SUMMARY:
This study is a 2-arm cluster randomized controlled trial with approximately 1,200 youth aged 14-19 years to assess the effectiveness of Yes and Know, a sexual health education program. To be eligible, participants must be 14-19 years old and English-speaking. Those in the treatment arm will receive Yes and Know, a synchronous virtual program delivered over multiple sessions totaling nine hours, along with asynchronous online activities and resources. Those in the control arm will receive a similarly structured program focused on nutrition education. Participants will complete brief online surveys at baseline and at 3 and 12 months after the synchronous sessions. The study will assess the program's effectiveness in reducing the prevalence of unprotected sex among youth and improving short-term outcomes, such as knowledge of reproductive health and healthy relationships, self-efficacy, and the use of reproductive health services.

DETAILED DESCRIPTION:
For the Yes and Know study, cohorts of 5-15 participants will be recruited and randomized into one of the two study conditions: Yes and Know: Life Skills intervention (intervention condition) or Yes and Know: Nutrition Skills intervention (comparison condition). The programs will be delivered by trained health educators through synchronous virtual sessions. Participants can access the supplemental resources and activities for their respective programs on the program's website. Each cohort will be recruited from a local partner site (with a focus on rural communities in the South and Southeast regions of the United States), and young people must have consent and provide their assent to be part of the study. Yes and Know: Sexual Health and Life Skills covers sexual and reproductive health, healthy relationships, life skills, and educational and career success. Yes and Know: Nutrition Skills covers learning to make healthy decisions about food, weight and disordered eating, and creating nourishing meals. Both programs consist of nine 60-minute synchronous group sessions, totaling nine hours, to be taught at least once a week (or more frequently depending on sites' scheduling).

ELIGIBILITY:
Inclusion Criteria:

* Ages 14-19; and
* English speaking.

Exclusion Criteria:

- Anyone not meeting inclusion criteria.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Rates of unprotected vaginal or anal sex | 12 months post-intervention
  Single measure constructed from the number of times had vaginal sex without a contraceptive method in the past 3 months; number of times had anal sex without a condom in the past 3 months.

SECONDARY OUTCOMES:
Use of sexual and reproductive health services in the past 3 months | 12 months post intervention
  Single dichotomous (yes/no) measure of whether the participant received any sexual or reproductive health services from a health care provider in the past 3 months, including condoms or other contraceptive methods, STI/HIV testing, prenatal care, or sexual health information.
Sexual and reproductive health knowledge | 3 months post intervention
  A measure of the % of correct answers (0% to 100%) on six survey questions that assess knowledge of sexual and reproductive health, developed for the study
Positive attitudes towards sexual consent | 3 months post intervention
  A measure comprised of 3 questions that assesses positive attitudes towards sexual consent.
  Scale scores range from 3 to 15 based on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree).
Self-efficacy in relationship communication | 3 months post intervention
  A measure comprised of 5 questions that assesses perceived self-efficacy in healthy relationship communication.
  Scale scores range from 5 to 25 based on a 5-point Likert scale (1 = not at all confident, 5=very confident).
Self-efficacy in using condoms correctly | 3 months post intervention
  A measure comprised of 3 questions that assesses perceived self-efficacy in using condoms correctly.
  Scale scores range from 3 to 12 based on a 4-point Likert scale (1 = no, definitely not, 4 = yes, definitely).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Braun, DrPH, MPH, Principal Investigator — ETR Associates; Karin K Coyle, PhD, Principal Investigator — ETR Associates
Locations (1):
- ETR Associates, Watsonville, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basen-Engquist K, Masse LC, Coyle K, Kirby D, Parcel GS, Banspach S, Nodora J. Validity of scales measuring the psychosocial determinants of HIV/STD-related risk behavior in adolescents. Health Educ Res. 1999 Feb;14(1):25-38. doi: 10.1093/her/14.1.25. PMID 10537945
- [Background] Humphreys TP, Brousseau MM. The sexual consent scale-revised: development, reliability, and preliminary validity. J Sex Res. 2010 Sep;47(5):420-8. doi: 10.1080/00224490903151358. PMID 19685367
- [Background] Scott, M.E., Moore, K.A., Fish, H., Benedetti, A., & Erikson, S. (2015). Healthy marriage and relationship education: Recommended outcome measures for adolescents. OPRE Report #2015-65a. Prepared by Child Trends. Washington, DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.